CLINICAL TRIAL: NCT00006484
Title: Randomized Phase III Trial Of Carboplatin And Paclitaxel Plus Tirapazamine Versus Carboplatin And Paclitaxel In Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy With or Without Tirapazamine in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068315; SWOG-S0003
Record Dates: First submitted 2000-11-06; First posted 2003-06-02 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2002-01

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Paclitaxel; Tirapazamine

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: tirapazamine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of carboplatin plus paclitaxel with or without tirapazamine in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of paclitaxel and carboplatin with or without tirapazamine on progression-free survival and overall survival in patients with stage IV and selected stage IIIB non-small cell lung cancer.
* Compare response rates in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to weight loss (less than 5% vs 5% or more), stage of disease (IIIB vs IV), and lactate dehydrogenase level (normal vs abnormal). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive tirapazamine IV over 2 hours followed by paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1.
* Arm II: Patients receive paclitaxel and carboplatin as in arm I. Treatment continues every 21 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for one year, and then every 6 months for 2 years, or until death.

PROJECTED ACCRUAL: Approximately 500 patients (250 per arm) will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven newly diagnosed advanced primary non-small cell lung cancer (NSCLC), including the following cellular types:

  * Adenocarcinoma
  * Large cell carcinoma
  * Squamous cell carcinoma
  * Unspecified carcinoma OR
* Recurrent disease after prior surgery and/or radiotherapy
* Stage IIIB disease

  * T4 lesion due to malignant pleural effusion OR
* Stage IV disease

  * Any T, any N, M1 (distant metastasis, including lesions in multiple lobes of the ipsilateral lung)
* Measurable or evaluable disease

  * Pleural effusions, ascites, and laboratory parameters not considered as only evidence of disease
  * Must be outside prior radiated field or area of prior surgical resection or new lesion must be present
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN

Renal:

* Creatinine no greater than ULN
* Creatinine clearance at least 50 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No peripheral neuropathy (motor or sensory) of grade 2 or greater
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I/II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for NSCLC

Chemotherapy:

* No prior systemic chemotherapy for NSCLC

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior thoracic or other major surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K. Williamson, MD, Study Chair — University of Kansas
Locations (93):
- United States (93):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Background] Lara PN Jr, Redman MW, Kelly K, Edelman MJ, Williamson SK, Crowley JJ, Gandara DR; Southwest Oncology Group. Disease control rate at 8 weeks predicts clinical benefit in advanced non-small-cell lung cancer: results from Southwest Oncology Group randomized trials. J Clin Oncol. 2008 Jan 20;26(3):463-7. doi: 10.1200/JCO.2007.13.0344. PMID 18202421
- [Background] Gandara DR, Kawaguchi T, Crowley JJ, et al.: Pharmacogenomic (PG) analysis of Japan-SWOG common arm study in advanced stage non-small cell lung cancer (NSCLC): a model for testing population-related pharmacogenomics. [Abstract] J Clin Oncol 25 (Suppl 18): A-7500, 2007.
- [Background] Lara PN Jr, Redman MW, Kelly K, et al.: Alternative measures predicting clinical benefit in advanced non-small cell lung cancer (NSCLC) from Southwest Oncology Group (SWOG) randomized trials: implications for clinical trial design. [Abstract] J Clin Oncol 24 (Suppl 18): A-7006, 365s, 2006.
- [Result] Mack PC, Redman MW, Chansky K, Williamson SK, Farneth NC, Lara PN Jr, Franklin WA, Le QT, Crowley JJ, Gandara DR; SWOG. Lower osteopontin plasma levels are associated with superior outcomes in advanced non-small-cell lung cancer patients receiving platinum-based chemotherapy: SWOG Study S0003. J Clin Oncol. 2008 Oct 10;26(29):4771-6. doi: 10.1200/JCO.2008.17.0662. Epub 2008 Sep 8. PMID 18779603
- [Result] Mack PC, Redman MW, Chansky K, et al.: Elevated osteopontin (OPN) plasma levels are highly prognostic in advanced non-small cell lung cancer (NSCLC): analysis of SWOG S0003. [Abstract] J Clin Oncol 24 (Suppl 18): A-7198, 413s, 2006.
- [Result] Williamson SK, Crowley JJ, Lara PN Jr, McCoy J, Lau DH, Tucker RW, Mills GM, Gandara DR; Southwest Oncology Group Trial S0003. Phase III trial of paclitaxel plus carboplatin with or without tirapazamine in advanced non-small-cell lung cancer: Southwest Oncology Group Trial S0003. J Clin Oncol. 2005 Dec 20;23(36):9097-104. doi: 10.1200/JCO.2005.01.3771. PMID 16361616
- [Result] Kimura T, Holland WS, Kawaguchi T, Williamson SK, Chansky K, Crowley JJ, Doroshow JH, Lenz HJ, Gandara DR, Gumerlock PH. Mutant DNA in plasma of lung cancer patients: potential for monitoring response to therapy. Ann N Y Acad Sci. 2004 Jun;1022:55-60. doi: 10.1196/annals.1318.010. PMID 15251940
- [Result] Williamson SK, Crowley JJ, Lara PN, et al.: S0003: paclitaxel/carboplatin (PC) versus PC + tirapazamine (PCT) in advanced non-small cell lung cancer (NSCLC). A phase III Southwest Oncology Group (SWOG) trial. [Abstract] Lung Cancer 41 (Suppl 2): A-O-89, S29, 2003.